CLINICAL TRIAL: NCT00163891
Title: A Prospective Randomised Two Month Trial Comparing Twho Chest Physiotherapy Protocols in Lung Transplant Recipients
Brief Title: Comparison of Two Chest Physiotherapy Protocols in Lung Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 107/03; A10503
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2005-09

CONDITIONS: Lung Transplantation
Keywords: Respiratory Therapy; Postoperative Care; Treatment Outcome

INTERVENTIONS:
Behavioral: Chest physiotherapy

SUMMARY:
Chest infection is a common complication following lung transplant (LTx). Chest physiotherapy is widely accepted as an integral part of the management of chest infections, however there is no evidence available regarding the effectiveness of chest physiotherapy regimes for LTx recipients.

There is no consensus regarding whether LTx recipients should be instructed to perform regular daily chest physiotherapy routines regardless of the presence of lung secretions (ie prophylatically) because of the changes in mucus clearance bought about by lung transplant, or only when they have a chest infection. Some clinicians believe that a prophylactic regimen may be beneficial.

This research will compare two chest physiotherapy treatment regimens - our current practice of chest physiotherapy during chest infections only (Treatment A) with an independently performed daily chest physiotherapy regimen regardless of the presence of a chest infection (Treatment B). From this research, we aim to develop evidence-based treatment guidelines.

DETAILED DESCRIPTION:
Very little is known about the effectiveness of chest physiotherapy protocols in lung transplant recipients. Clinical practice is based upon the experiences of individual clinicians and generalisations from other patient populations.

There is anecdotal evidence (from discussion with physiotherapists at the European Cystic Fibrosis Conference, 2001) that some lung transplant centres are advising their patients to undertake daily (prophylactic) chest physiotherapy as part of their usual routine. They believe that this may compensate for the reduced stimulus to cough caused by the lack of vagal nerve supply to the transplanted lung/s.There is no evidence that this time consuming intervention is of any benefit to the patient in the short or longer term.

Some patients have bronchial anastomotic complications and dynamic airway collapse that may further impair secretion removal. The mechanical effects of Positive Expiratory Pressure (PEP) mask Physiotherapy, particularly its ability to splint open airways, provides a theoretical basis for why this technique may be beneficial to lung transplant recipients. We have also noted a clinical benefit in a small number of patients who have been treated with PEP.

This study aims to evaluate two chest physiotherapy protocols using a variety of outcome measures and act as a starting point for future/ongoing research in this important clinical area.

This study is a prospective randomised two month trail comparing two chest physiotherapy protocols in lung transplant recipients.

The protocols are:

Treatment A - Positive expiratory pressure (PEP) mask physiotherapy in upright sitting carried out only during chest infections

Treatment B - Positive expiratory pressure (PEP) mask physiotherapy in upright sitting performed twice daily as a prophylactic routine

The null hypotheses are:

1. Comparing Treatment A & B, there will be no difference in:

   * Lung function
   * Chest X ray (Brasfield scores)
   * Airway status (Bronchoscopy scores)
   * Days in hospital due to chest infection
   * Days on antibiotics
   * Exercise capacity (6 minute walk test)
   * Quality of life
2. There will be no difference in patient adherence to the alternative protocols.
3. There will be no difference in patient satisfaction with the alternative protocols.

ELIGIBILITY:
Inclusion Criteria:

* All lung transplant recipients treated at The Alfred will be invited to participate in the study at three weeks following lung transplantation.

Exclusion Criteria:

* ventilator dependent
* tracheostomy insitu
* pneumothorax
* major myopathy
* oxygen requirement of greater than 4 litres per minute
* or any condition that prevents them from performing PEP mask chest physiotherapy at the time of recruitment to the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-09

PRIMARY OUTCOMES:
Lung function
Chest radiographic score -Brasfield Score
Bronchoscopy score
Days in hospital due to chest infection
Antibiotic use
Quality of Life - SF-36 Health Survey
Functional exercise capacity - 6 minute walk test

SECONDARY OUTCOMES:
Patient adherence to the alternative protocols
Patient satisfaction with the alternative protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bailey, M Stat PhD, Principal Investigator — Dept of Epidemiology & Preventative Medicine Monash University; Prue E Munro, B Physio GradDip HealthMan, Principal Investigator — The Alfred; Brenda B Button, DPhysio PhD, Principal Investigator — The Alfred; Samantha Ellis, Principal Investigator — The Alfred; Greg I Snell, MBBS FRACP, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia